CLINICAL TRIAL: NCT06389721
Title: Understanding and Preventing Cortical Mechanisms of Chemotherapy-induced Peripheral Neuropathy
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0145; NCI-2024-03672 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Participants in Group 1, you will have an EEG and complete one questionnaire prior to your first dose of chemotherapy and once monthly until the end of your chemotherapy (for a maximum of 6 measurements).
  Interventions: Diagnostic Test: Electroencephalogram (EEG)
- Cohort 2: Participants in Group 2, you will have an EEG, and complete a questionnaire before and after your chemotherapy regimen. Participants will also have a treatment called closed-loop brain-computer interface (clBCI) training twice a week for the 2 weeks leading up to starting chemotherapy, and then twice a week during chemotherapy, for a maximum of 32 sessions, which you will be able to do at home.
  Interventions: Diagnostic Test: Electroencephalogram (EEG)

INTERVENTIONS:
Diagnostic Test: Electroencephalogram (EEG) — Measure the electrical activity of your brain before you receive chemotherapy treatment and once monthly for a maximum of 6 measurements.

SUMMARY:
Cohort 1: To track the onset and progression of a condition called chemotherapy-induced peripheral neuropathy (CIPN).

Cohort 2: To track the onset and progression of a condition called chemotherapy-induced peripheral neuropathy (CIPN) and to test a certain type of experimental neuromodulation (stimulation of the brain) with a device called a closed-loop brain-computer interface (clBCI) to see if can help to prevent pain due to CIPN.

DETAILED DESCRIPTION:
Primary Objectives:

Objective 1 (Primary Objective): to examine preliminary baseline and serial electrophysiological markers associated with the onset and development of CIPN by tracking brain activity and CIPN symptoms throughout chemotherapy treatment.

Secondary Objectives:

Objective 2 (Secondary Objective): To preliminarily evaluate whether a clBCI program can regulate changes in EEG that are associated with CIPN while participants are undergoing chemotherapy.

Exploratory Objective: Explore whether there are associations between change in brain function and subjective report of CIPN.

ELIGIBILITY:
Inclusion criteria:

Objective 1 Inclusion criteria

1. Participants must have the ability to understand and read English, sign a written informed consent, and be willing to follow protocol requirements.
2. ECOG Performance Status of 0-2;
3. Willing to come to MD Anderson for the imaging sessions.
4. Are 18 years of age or above.
5. Have a diagnosis of breast cancer.
6. will receive chemotherapy including doxorubicin, cyclophosphamide, docetaxel, or paclitaxel;

Objective 2 Inclusion criteria:

1) Inclusion criteria: Identical to Objective 1 and are willing to participate in the therapy sessions at their homes.

Exclusion Criteria

Objective 1 Exclusion criteria:

1. Participants who are taking any antipsychotic medications.
2. With active CNS disease, such as clinically evident metastases or leptomeningeal disease, dementia, or encephalopathy.
3. Have ever been diagnosed with bipolar disorder or schizophrenia.
4. Known, previously diagnosed peripheral neuropathy from causes other than chemotherapy; and
5. A history of head injury or who have known seizure activity, or with a prior history of chemotherapy.
6. Patients who will be administered ddAC->T.

Objective 2 Exclusion criteria

1) Same exclusion criteria as in Objective1. Medication usage will be tracked for patients in all groups. Once prescribed, participants must remain on a stable course of medications throughout the course of chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants at MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Prinsloo, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org